CLINICAL TRIAL: NCT05999201
Title: Effect of Craniocervical Neural Mobilization on Quality of Life in Patients With Primary Tension Headache
Acronym: TTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdul Hamid Elgendy, principle investigator amira mohamed abdul hamid, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003179
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Tension-Type Headache
Keywords: craniocervical neural mobilization; quality of life; primary tension headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Intervention Model Description: Craniocervical Neural Mobilization and selected physiotherapy program
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- craniocervical neural mobilization (Experimental): the patients will receive craniocervical neural mobilization and a selected physiotherapy program twice a week for four weeks
  Interventions: Other: craniocervical neural mobilization; Other: selected physiotherapy program
- selected physiotherapy program (Active Comparator): the patients will receive a selected physiotherapy program twice a week for four weeks
  Interventions: Other: selected physiotherapy program

INTERVENTIONS:
Other: craniocervical neural mobilization — the patients will receive The craniocervical neural mobilization in the form of passive craniocervical flexion in which An anterior rotation of the head will be done which stimulates the meninges.To increase mechanical stress in the nervous system, patients will be asked to do a descent and retropulsion of the shoulders while gradually extending both elbows. in addition to Passive lateral cervical sliding and Craniocervical flexion with mouth opening.The neural mobilization should be mild, progressive, and slow. The protocol lasted 15 minutes and also the patients will receive selected physiotherapy program
  Arms: craniocervical neural mobilization
Other: selected physiotherapy program — the patients will receive selected physiotherapy program in the form of Suboccibital muscles inhibition suboccipital inhibition technique (SIT), from supine lying position, the therapist will sit at the patient's head head with the elbows rested on the surface of the table. Then, the therapist will place both hands behind the head of the patient with the palms facing upwards, the fingers flexed, and the finger pads positioned on the posterior arch of the atlas to allow the occiput to rest in the palm of the hands. the patients will receive also trigger point release technique in the form of An ischemic compression for sternocleidomastoid muscle, temporal muscle, upper trapezius muscle and splines muscles

SUMMARY:
this study will be conducted to investigate the effect of craniocervical neural mobilization on quality of life in patients with primary tension headache.

DETAILED DESCRIPTION:
The World Health Organization estimates that the three most prevalent neurologic disorders worldwide are tension-type headache (1.5 billion), migraine (958.8 million), and medication overuse headache (58.5 million). Collectively, these three disorders contribute approximately 17% to the global burden of neurologic diseases, with migraine the second most disabling disease overall. TTH (Tension Type of Headache) is defined as mild to moderate band-like pressure headache with few associated symptoms. It varies considerably in frequency and duration, from rare, short-lasting episodes of discomfort to frequent, long-lasting, or even continuous disabling headaches.Physiotherapy treatment based on manual therapy achieved positive outcomes in pain intensity and frequency, disability, impact of headache, quality of life, and craniocervical range of motion in adults with TTH. Although pervious findings showed a clinical improvement, there is no clear evidence that one technique is superior to another.Neurodynamic techniques can improve mechanical functions in nerve structures, such as tension and sliding functions. When the nerve structure experiences clamping and disrupts mobility, pain occurs along the nerve. Neurodynamic sliding techniques play a major role in improving blood circulation and axonal transport, as well as increasing nerve integrity and reducing the pressure caused by intraneural and extraneural fibrosis. thirty patients with tension headache will be allocated randomly into two equal groups. the first one will receive craniocervical mobilization and a selected physiotherapy program and the control group will receive selected physiotherapy program for one month.

ELIGIBILITY:
Inclusion Criteria:

* The type of headache will be primary tension type of headache.
* Age of subjects will range from 25-40 years.
* The duration of headaches swill be one years ago.
* Body mass index from 25 to less than 30.

Exclusion Criteria:

* Major neurological conditions (e.g. stroke, multiple sclerosis, epilepsy, brain tumor, meningitis, and hypertension).
* Patients with cervical spinal cord injury, recent trauma of head.
* Patients with auditory and visual impairments.
* Smoker and addicted subjects.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
life disability | up to four weeks
  Headache Impact Test-6 scale will be used to assess life disability.It is a six-item, self-report, retrospective questionnaire. The six items in the HIT-6 address such aspects of quality of life as pain, social functioning, cognitive functioning, and psychological distress.The HIT-6 is scored by giving these responses a value of 6, 8, 10, 11, and 13, respectively. The four headache impact severity categories are little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78).
frequency and severity of headache | up to four weeks
  headache disability index will be used to assess the frequency and severity of headache. The questionnaire begins with two items that assess pain severity (mild, moderate, and severe) and frequency (once month, from 1 to 4 times a month, and more than once a week). It also includes 25 question on functional sub-scale (12 items) and emotional subscale (13 items) with three possible response option (No=0 points; Sometimes=2 points; Yes=4 points). The maximum score is 100 points, ranging from 0=no disability to 100=severe disability. A total score of 10-28 is considered o indicate mild disability; 30-48 is moderate disability; 50-68 is sever disability; 72 or more is complete disability
pain intensity | up to four weeks
  visaul analogue scale will be used to assess pain intensity. Patients will be informed about visual analog scale that has two ends ; 0: no pain; 10: maximum pain.